CLINICAL TRIAL: NCT00805220
Title: Nordic Walking for Frail Elderly: a Randomized Pilot Trial
Brief Title: Nordic Walking as Gait Training for Frail Elderly
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: McGill University (Other)
Responsible Party: Nancy E. Mayo, BSc(PT), MSc, PhD, McGill University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NWS-001
Record Dates: First submitted 2008-12-08; First posted 2008-12-09 (Estimated); Last update posted 2009-09-02 (Estimated); Status verified 2009-09

CONDITIONS: Frail Elderly
Keywords: frail elderly walking capacity walk training Nordic Walking
MeSH Terms: interventions — Nordic Walking

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Regular overground walking without poles
  Interventions: Other: Nordic Walking
- 2 (Experimental): Nordic Walking
  Interventions: Other: Nordic Walking

INTERVENTIONS:
Other: Nordic Walking — Walking training with and without poles will be twice a week. The sessions last 20 minutes each and consist of walking, stretching and mobility exercises. This will last 8 weeks in a total of 16 sessions. A therapist will closely monitor your exercises and modify them according to your needs and comfort
  Other Names: PoleStriding; Exerstriding

SUMMARY:
The elderly are the fastest growing proportion of the population. Ageism implies a decline of physical functions affecting functional and safe ambulation. Based on the ICF model intervening in walking capacity could have favourable impact on quality of life of frail elders. Over ground walking training is indicated as a possible exercise. However, to achieve positive results on walking capacity, an exercise-dose response is needed. A more intensive way of promoting walking training is to add skiing poles while walking, a technique called Nordic Walking (NW). This study will be the first to compare NW with usual walking training. It aims to estimate for frail elderly the relative efficacy in improving functional walking capacity of two gait training strategies: NW and usual walking training and explore its impact on fear of falling. This study hypothesized that participants receiving Nordic Walking will walk longer, faster and fear less. NW if proven effective will positively impact on the functional capacities and quality of life of frail elders and provide an more intense method of walking training.

DETAILED DESCRIPTION:
This is a single blind, randomized, pilot trial designed to estimate the amount of change between two programs. Subjects will be randomized and stratified by setting into one of two groups, over ground walking training with poles (Nordic Walking) or traditional over ground walking training (without poles). Randomization will be computer generated using randomization scheme from the website Randomization.com at http://www.randomization.com Basic descriptive statistics will be used to characterize the participants and compare the two groups at baseline. Paired t-test will be used to estimate the efficacy of each intervention. Effects size of each interventions and its ratio will be calculated. Group-specific change score will be calculated to explore the impact of prognostic variables (age, gender, number of comorbities, baseline gait speed) on change of an outcome (with or without poles).

ELIGIBILITY:
Inclusion Criteria:

1. 65 years old or more
2. undergoing rehabilitation program or living a residence facility
3. medically stable or in their usually state of health.

Exclusion Criteria:

1. severe cognitive impairments (short mini mental score less than 14/18)47
2. unable to ambulate a minimum of 15 meters with or without aids
3. without mobility restrictions as represented by a gait speed greater than 1.2 m/s
4. moderate to severe limitations of upper extremity represented by a shoulder flexion range of motion (ROM) less than 90 degrees and extension less than 20 degrees; elbow flexion ROM less than 90 degrees; and with a poor grip judged by the ability to release a can of 5 cm diameter
5. pathological or musculoskeletal conditions of the upper extremity
6. individuals unable to attend a minimum of eight weeks of intervention.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2008-12; Primary Completion 2009-06 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
6 Minute Walk Test 5 Meter Walk Test Activities-Specific Balance Confidence (ABC) Scale | Baseline, 3 weeks follow-up, 8 weeks follow-up

SECONDARY OUTCOMES:
Berg Balance Scale; CHAMPS; Lower Extremity Functional Scale; Visual Analogue Scale of Pain; EuroQol 5D. | Baseline, 3 weeks follow-up, 8 weeks follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Mayo, BSc MSc PhD, Principal Investigator — McGill University
Locations (2):
- Canada (2):
  - Geriatric Day Hospital (GDH) at the Royal Victoria Hospital (RVH), Montreal, Quebec
  - Richardson Hospital, Montreal, Quebec

REFERENCES:
- [Derived] Figueiredo S, Finch L, Mai J, Ahmed S, Huang A, Mayo NE. Nordic walking for geriatric rehabilitation: a randomized pilot trial. Disabil Rehabil. 2013 Jun;35(12):968-75. doi: 10.3109/09638288.2012.717580. Epub 2012 Oct 15. PMID 23066879
- See also: Pete Edwards and The American Nordic Walking System — http://www.skiwalking.com